CLINICAL TRIAL: NCT02730169
Title: A Phase IIb Multicentre, Double-Blind, Dose-Ranging, Randomised, Placebo-Controlled Study Evaluating Safety and Efficacy of BGS649 in Male Obese Subjects With Hypogonadotropic Hypogonadism
Brief Title: Safety and Efficacy of BGS649 in Male Obese Subjects With Hypogonadotropic Hypogonadism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mereo BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MBGS205
Record Dates: First submitted 2016-03-17; First posted 2016-04-06 (Estimated); Results first posted 2020-11-25 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-08

CONDITIONS: Hypogonadotropic Hypogonadism
Keywords: Hypogonadotropic; hypogonadism; testosterone
MeSH Terms: conditions — Hypogonadism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- BGS649 0.1 mg (Experimental): BGS649 0.1 mg weekly (1 BGS649 0.1 mg capsule and 2 indistinguishable placebo capsules)
  Interventions: Drug: BGS649
- BGS649 0.3 mg (Experimental): BGS649 0.3 mg weekly (3 BGS649 0.1 mg capsules)
  Interventions: Drug: BGS649
- BGS649 1.0 mg (Experimental): BGS649 1.0 mg weekly (1 BGS649 1.0 mg capsule and 2 indistinguishable placebo capsules)
  Interventions: Drug: BGS649
- Placebo (Placebo Comparator): Placebo weekly (3 indistinguishable placebo capsules)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BGS649 — Capsules were taken weekly for a maximum of 24 weeks
  Arms: BGS649 0.1 mg; BGS649 0.3 mg; BGS649 1.0 mg
Drug: Placebo — Capsules were taken weekly for a maximum of 24 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of BGS649 in male obese subjects with hypogonadotropic hypogonadism. All subjects will be treated for a maximum of 24 weeks. Some subjects who complete 24 weeks of treatment will be invited to participate in a 6-month blinded safety extension study (Protocol MBGS206). The study is planned to enroll 268 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Adult male subject aged 18 to 65 years inclusive
* BMI > 30 kg/m2 and < 50 kg/m2
* Serum total testosterone concentration below the normal range
* LH levels below the upper limit of normal
* Oestradiol levels within or above the normal range of approved assay
* At least two symptoms of androgen deficiency present for at least 2 months prior to the first Screening Visit, with at least one of these being a sexual dysfunction

Exclusion Criteria:

* Evidence of clinically significant endocrinopathy at screening that may interfere with the study assessments
* Other types of hypogonadotropic hypogonadism or primary hypogonadism
* Any other pituitary or hypothalamic disease

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2016-05-12 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Jones, Principal Investigator — Barnsley Hospital NHS Foundation Trust
Locations (63):
- United States (48):
  - Mereo Research Site, Birmingham, Alabama
  - Mereo Research Site, Mobile, Alabama
  - Mereo Research Site, Chandler, Arizona
  - Mereo Research Site, Phoenix, Arizona
  - Mereo Research Site, Scottsdale, Arizona
  - Mereo Research Site, Anaheim, California
  - Mereo Research Site, Carlsbad, California
  - Mereo Research Site, Greenbrae, California
  - Mereo Research Site, Lincoln, California
  - Mereo Research Site, Los Angeles, California
  - Mereo Research Site, San Diego, California
  - Mereo Research Site, Bradenton, Florida
  - Mereo Research Site, DeLand, Florida
  - Mereo Research Site, Fort Myers, Florida
  - Mereo Research Site, Hialeah, Florida
  - Mereo Research Site, Homestead, Florida
  - Mereo Research Site, St. Petersburg, Florida
  - Mereo Research Site, Meridian, Idaho
  - Mereo Research Site, Gurnee, Illinois
  - Mereo Research Site, Evansville, Indiana
  - Mereo Research Site, New Orleans, Louisiana
  - Mereo Research Site, Baltimore, Maryland
  - Mereo Research Site, Elkridge, Maryland
  - Mereo Research Site, St Louis, Missouri
  - Mereo Research Site, Omaha, Nebraska
  - Mereo Research Site, Henderson, Nevada
  - Mereo Research Site, Las Vegas, Nevada
  - Mereo Research Site, Albany, New York
  - Mereo Research Site, Garden City, New York
  - Mereo Research Site, Great Neck, New York
  - Mereo Research Site, New York, New York
  - Mereo Research Site, Rochester, New York
  - Mereo Research Site, Charlotte, North Carolina
  - Mereo Research Site, Raleigh, North Carolina
  - Mereo Research Site, Winston-Salem, North Carolina
  - Mereo Research Site, Middleburg Heights, Ohio
  - Mereo Research Site, Mt. Pleasant, South Carolina
  - Mereo Research Site, Nashville, Tennessee
  - Mereo Research Site, Smyrna, Tennessee
  - Mereo Research Site, Spring Hill, Tennessee
  - Mereo Research Site, Dallas, Texas
  - Mereo Research Site, Fort Worth, Texas
  - Mereo Research Site, Pearland, Texas
  - Mereo Research Site, San Antonio, Texas
  - Mereo Research Site, Murray, Utah
  - Mereo Research Site, West Jordan, Utah
  - Mereo Research Site, Norfolk, Virginia
  - Mereo Research Site, Kenosha, Wisconsin
- Italy (4):
  - Mereo Research Site, Ancona
  - Mereo Research Site, Parma
  - Mereo Research Site, Roma
  - Mereo Research Site, Siena
- Spain (4):
  - Mereo Research Site, Coslada
  - Mereo Research Site, Girona
  - Mereo Research Site, Madrid
  - Mereo Research Site, Majadahonda
- United Kingdom (7):
  - Mereo Research Site, Barnsley
  - Mereo Research Site, Coventry
  - Mereo Research Site, Dundee
  - Mereo Research Site, Edinburgh
  - Mereo Research Site, Hull
  - Mereo Research Site, Manchester
  - Mereo Research Site, Newcastle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jones TH, Dobs AS, Randeva H, Moore W, Parkin JM. Leflutrozole in male obesity-associated hypogonadotropic hypogonadism: Ph 2b double-blind randomised controlled trial. Eur J Endocrinol. 2023 Sep 1;189(3):297-308. doi: 10.1093/ejendo/lvad099. PMID 37579053

RESULTS

PARTICIPANT FLOW:
Groups:
- BGS649 0.1 mg: BGS649 0.1 mg weekly (1 BGS649 0.1 mg capsule and 2 indistinguishable placebo capsules)
  BGS649: Capsules will be taken weekly for a maximum of 24 weeks
- BGS649 0.3 mg: BGS649 0.3 mg weekly (3 BGS649 0.1 mg capsules)
  BGS649: Capsules will be taken weekly for a maximum of 24 weeks
- BGS649 1.0 mg: BGS649 1.0 mg weekly (1 BGS649 1.0 mg capsule and 2 indistinguishable placebo capsules)
  BGS649: Capsules will be taken weekly for a maximum of 24 weeks
- Placebo: Placebo weekly (3 indistinguishable placebo capsules)
  Placebo: Capsules will be taken weekly for a maximum of 24 weeks
Period: Overall Study
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg | Placebo
Started | 67 | 66 | 67 | 71
Completed | 53 | 45 | 50 | 55
Not Completed | 14 | 21 | 17 | 16
Not completed — Protocol Violation | 1 | 0 | 0 | 1
Not completed — Adverse Event | 2 | 3 | 3 | 0
Not completed — Adverse Event of Special Interest | 0 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 6 | 11 | 6 | 8
Not completed — Lost to Follow-up | 5 | 6 | 5 | 6
Not completed — Other | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg | Placebo | Total
Number analyzed (Participants) | 67 | 66 | 67 | 71 | 271
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (8.39) | 51.6 (7.31) | 49.6 (9.72) | 50.9 (9.17) | 50.8 (8.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 67 | 66 | 67 | 71 | 271
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race as defined by the NIH/OMB guidelines
  Participants
    American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
    Asian | 0 | 2 | 2 | 0 | 4
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
    Black or African American | 12 | 13 | 15 | 7 | 47
    White | 53 | 49 | 49 | 61 | 212
    More than one race | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 1 | 2 | 0 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Normalised Testosterone After 24 Weeks of Study Treatment
Description: Percentage of patients with normalised testosterone i.e. testosterone in the range 300-1000ng/dL after 24 weeks of study treatment. The primary objective was considered met, if greater than or equal to 75% of the participants in any arm normalised.
Time Frame: 24 weeks of treatment
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg | Placebo
Number analyzed (Participants) | 67 | 65 | 67 | 71
Participants | 59 | 62 | 63 | 7

2. Secondary Outcome: The Proportion of Subjects That Have Normalization of Total Testosterone Serum Concentrations From Baseline to Week 24
Description: Normalised total testosterone level was defined as between 300-1000 ng/dL (10.4-35 nmol/L) inclusive. Levels >1000 ng/dL were considered super-physiological outside the normal range.
Time Frame: Baseline, Day 8, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks and 24 weeks
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg | Placebo
Number analyzed (Participants) | 67 | 65 | 67 | 71
Participants
  Baseline | 7 | 12 | 11 | 7
  Visit 2 (Day 8): number analyzed (Participants) | 67 | 62 | 64 | 68
  Visit 2 (Day 8) | 54 | 53 | 57 | 7
  Visit 3 (Week 4): number analyzed (Participants) | 67 | 65 | 66 | 71
  Visit 3 (Week 4) | 63 | 62 | 64 | 10
  Visit 4 (Week 8) | 63 | 61 | 65 | 11
  Visit 5 (Week 12) | 58 | 62 | 64 | 7
  Visit 6 (Week 16) | 57 | 63 | 63 | 8
  Visit 7 (Week 20) | 57 | 63 | 66 | 9
  Visit 8 (Week 24) | 59 | 62 | 63 | 7

3. Secondary Outcome: Proportion of Subjects That Overshoot Testosterone (Total Testosterone Above 1000 ng/dL [35 Nmol/L]) From Baseline to Week 24
Description: Testosterone overshoot was defined as total testosterone above 1000 ng/dL (35 nmol/L). Samples were collected in the morning before 11 am pre dose.
Time Frame: Baseline, Day 8, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks and 24 weeks
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg | Placebo
Number analyzed (Participants) | 67 | 65 | 67 | 71
Participants
  Baseline | 0 | 0 | 0 | 0
  Visit 2 (Day 8): number analyzed (Participants) | 67 | 61 | 64 | 68
  Visit 2 (Day 8) | 0 | 0 | 0 | 0
  Visit 3 (Week 4): number analyzed (Participants) | 66 | 60 | 63 | 65
  Visit 3 (Week 4) | 0 | 0 | 0 | 0
  Visit 4 (Week 8): number analyzed (Participants) | 62 | 59 | 57 | 66
  Visit 4 (Week 8) | 0 | 0 | 1 | 0
  Visit 5 (Week 12): number analyzed (Participants) | 56 | 53 | 53 | 60
  Visit 5 (Week 12) | 0 | 0 | 2 | 2
  Visit 6 (Week 16): number analyzed (Participants) | 54 | 50 | 50 | 55
  Visit 6 (Week 16) | 0 | 0 | 2 | 1
  Visit 7 (Week 20): number analyzed (Participants) | 52 | 43 | 46 | 55
  Visit 7 (Week 20) | 0 | 0 | 0 | 1
  Visit 8 (Week 24): number analyzed (Participants) | 52 | 40 | 39 | 51
  Visit 8 (Week 24) | 0 | 0 | 1 | 0

4. Secondary Outcome: Normalization of Total Testosterone Serum Concentrations in ≥ 90% Subjects After 24 Weeks of Treatment.
Description: Normalized total testosterone level was defined as between 300-1000 ng/dL (10.4-35 nmol/L) inclusive. Levels >1000 ng/dL were considered super-physiological outside the normal range. This secondary outcome measure was considered to have been met for a dose if ≥ 90% of subjects in the intent-to-treat (ITT) population had normalisation of total testosterone levels at Week 24.
Time Frame: 24 weeks of treatment
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg | Placebo
Number analyzed (Participants) | 67 | 65 | 67 | 71
Participants | 59 | 62 | 63 | 7

5. Secondary Outcome: Mean (SD) Change From Baseline in Luteinizing Hormone (LH) to Week 24.
Description: LH was measured at screening, baseline. The Baseline was defined as the last non-missing value collected before the first study treatment administration, including unscheduled assessments.
Time Frame: Day 8, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks and 24 weeks
Population: ITT Population
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg | Placebo
Number analyzed (Participants) | 67 | 65 | 67 | 71
mIU/mL
  Visit 2 (Day 8): number analyzed (Participants) | 67 | 62 | 64 | 70
  Visit 2 (Day 8) | 1.680 (1.7503) | 2.095 (1.3719) | 3.309 (1.8200) | -0.183 (1.3531)
  Visit 3 (Week 4): number analyzed (Participants) | 66 | 63 | 64 | 67
  Visit 3 (Week 4) | 2.237 (2.1982) | 3.626 (2.6519) | 5.235 (4.8684) | -0.385 (1.2423)
  Visit 4 (Week 8): number analyzed (Participants) | 62 | 58 | 57 | 65
  Visit 4 (Week 8) | 2.272 (2.1908) | 3.653 (3.0907) | 5.676 (4.1471) | -0.169 (1.5237)
  Visit 5 (Week 12): number analyzed (Participants) | 58 | 55 | 55 | 62
  Visit 5 (Week 12) | 2.503 (2.2230) | 3.511 (3.7050) | 5.064 (3.9739) | -0.341 (1.4575)
  Visit 6 (Week 16): number analyzed (Participants) | 54 | 50 | 52 | 58
  Visit 6 (Week 16) | 2.557 (1.6964) | 3.704 (3.6269) | 5.004 (4.3397) | -0.395 (1.4793)
  Visit 7 (Week 20): number analyzed (Participants) | 53 | 45 | 48 | 56
  Visit 7 (Week 20) | 2.553 (2.2380) | 3.653 (3.7381) | 4.884 (3.9297) | -0.193 (1.3585)
  Visit 8 (Week 24): number analyzed (Participants) | 52 | 41 | 42 | 54
  Visit 8 (Week 24) | 2.108 (1.9892) | 3.560 (3.6138) | 5.209 (4.4894) | -0.043 (1.5575)

6. Secondary Outcome: Mean (SD) Change From Baseline in Follicle Stimulating Hormone (FSH) to Week 24.
Description: FSH was measured at baseline, Visit 1 through 8 and follow-up. Baseline was defined as the last non-missing value collected before the first study treatment administration, including unscheduled assessments.
Time Frame: Day 8, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks and 24 weeks
Population: ITT Population
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg | Placebo
Number analyzed (Participants) | 67 | 65 | 66 | 69
mIU/mL
  Visit 2 (Day 8): number analyzed (Participants) | 66 | 62 | 63 | 68
  Visit 2 (Day 8) | 3.553 (2.2022) | 4.575 (2.0756) | 5.307 (2.8315) | -0.51 (0.8273)
  Visit 3 (Week 4): number analyzed (Participants) | 65 | 63 | 63 | 64
  Visit 3 (Week 4) | 4.158 (2.1353) | 5.540 (2.8344) | 6.551 (4.2155) | -0.111 (1.0638)
  Visit 4 (Week 8): number analyzed (Participants) | 61 | 58 | 57 | 63
  Visit 4 (Week 8) | 4.318 (2.4147) | 5.878 (2.9916) | 7.620 (4.7883) | 0.047 (1.2241)
  Visit 5 (Week 12): number analyzed (Participants) | 57 | 55 | 54 | 60
  Visit 5 (Week 12) | 4.809 (2.5582) | 5.768 (3.2474) | 8.132 (5.9526) | -0.075 (1.0723)
  Visit 6 (Week 16): number analyzed (Participants) | 53 | 50 | 52 | 56
  Visit 6 (Week 16) | 5.188 (2.6876) | 6.350 (3.4261) | 8.045 (6.1773) | -0.165 (1.1924)
  Visit 7 (Week 20): number analyzed (Participants) | 52 | 45 | 48 | 54
  Visit 7 (Week 20) | 5.059 (2.5714) | 6.073 (3.5199) | 8.409 (6.6502) | -0.030 (1.0932)
  Visit 8 (Week 24): number analyzed (Participants) | 51 | 41 | 42 | 52
  Visit 8 (Week 24) | 4.836 (2.6901) | 6.183 (3.4817) | 8.282 (7.0523) | 0.038 (1.2164)

7. Secondary Outcome: Descriptive Summary (Geometric Mean [95% CI]) of BGS649 Plasma PK Concentration Values to 24 Weeks.
Description: Plasma PK sampling for BGS649 was performed at Weeks 12 and 24. BGS649 PK plasma concentrations were summarised for the PK population by descriptive statistics.
Time Frame: Week 12 (pre-dose and 1 hour post-dose), week 24 and week 24/End of treatment
Population: PK population
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg
Number analyzed (Participants) | 64 | 59 | 65
ng/mL
  Visit 5 (Week 12), Pre-Dose: number analyzed (Participants) | 54 | 51 | 53
  Visit 5 (Week 12), Pre-Dose | 0.73 [0.64 to 0.83] | 2.55 [2.33 to 2.80] | 8.93 [8.29 to 9.62]
  Visit 5 (Week 12), 1 hour Post-Dose: number analyzed (Participants) | 55 | 51 | 52
  Visit 5 (Week 12), 1 hour Post-Dose | 1.43 [1.24 to 1.65] | 4.39 [3.89 to 4.97] | 14.91 [13.52 to 16.45]
  Visit 8 (Week 24): number analyzed (Participants) | 47 | 36 | 41
  Visit 8 (Week 24) | 0.85 [0.72 to 1.00] | 2.97 [2.20 to 4.00] | 10.04 [8.23 to 12.25]
  Visit 8 (Week 24)/End of Treatment: number analyzed (Participants) | 51 | 43 | 51
  Visit 8 (Week 24)/End of Treatment | 0.78 [0.64 to 0.97] | 2.76 [2.14 to 3.57] | 9.10 [7.61 to 10.89]

8. Secondary Outcome: Descriptive Summary (Geometric Mean [95% CI]) of BGS649 Semen PK Concentration Values at 24 Weeks.
Description: Semen PK sampling for BGS649 was performed at Visit 8 (End of Treatment). BGS649 PK semen concentrations were summarised for the PK population by descriptive statistics.
Time Frame: Week 24 and week 24/End of treatment
Population: PK population
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg
Number analyzed (Participants) | 64 | 59 | 65
ng/mL
  Visit 8 (Week 24): number analyzed (Participants) | 22 | 13 | 15
  Visit 8 (Week 24) | 0.51 [0.43 to 0.61] | 1.95 [1.60 to 2.38] | 5.81 [4.63 to 7.28]
  Visit 8 (Week 24)/End of Treatment: number analyzed (Participants) | 25 | 17 | 18
  Visit 8 (Week 24)/End of Treatment | 0.49 [0.42 to 0.58] | 1.58 [1.19 to 2.08] | 5.28 [4.16 to 6.71]

9. Other Pre Specified Outcome: Mean (SD) Change From Baseline in Prostate Specific Antigen (PSA) to Week 24.
Description: PSA was measured alongside other clinical chemistry parameters at screening, baseline, Visits 1 through 8 and at follow-up.
Time Frame: Baseline, Day 8, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks and 24 weeks
Population: Safety Population
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg | Placebo
Number analyzed (Participants) | 67 | 66 | 67 | 71
ug/L
  Visit 2 (Day 8): number analyzed (Participants) | 67 | 62 | 64 | 70
  Visit 2 (Day 8) | 0.045 (0.1840) | 0.040 (0.4830) | 0.011 (0.4606) | 0.015 (0.2179)
  Visit 3 (Week 4): number analyzed (Participants) | 66 | 63 | 64 | 67
  Visit 3 (Week 4) | 0.141 (0.1742) | 0.082 (0.5198) | 0.092 (0.4338) | 0.038 (0.2700)
  Visit 4 (Week 8): number analyzed (Participants) | 62 | 59 | 59 | 66
  Visit 4 (Week 8) | 0.166 (0.2651) | 0.105 (0.4747) | 0.132 (0.3343) | 0.055 (0.4500)
  Visit 5 (Week 12): number analyzed (Participants) | 58 | 55 | 54 | 62
  Visit 5 (Week 12) | 0.190 (0.3895) | 0.271 (0.9626) | 0.178 (0.5405) | 0.039 (0.4382)
  Visit 6 (Week 16): number analyzed (Participants) | 53 | 51 | 52 | 58
  Visit 6 (Week 16) | 0.147 (0.2655) | 0.102 (0.5500) | 0.160 (0.4037) | 0.016 (0.2631)
  Visit 7 (Week 20): number analyzed (Participants) | 53 | 45 | 48 | 56
  Visit 7 (Week 20) | 0.158 (0.2913) | 0.480 (2.6029) | 0.116 (0.4560) | 0.022 (0.3942)
  Visit 8 (Week 24): number analyzed (Participants) | 52 | 40 | 42 | 55
  Visit 8 (Week 24) | 0.218 (0.4312) | 0.391 (1.8627) | 0.085 (0.2930) | 0.067 (0.4787)

10. Other Pre Specified Outcome: Mean (SD) Change From Baseline in Haematocrit to Week 24.
Description: Haematocrit was measured alongside other haematology parameters at screening, baseline, Visits 1 through 8 and at follow-up.
Time Frame: Day 8, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks and 24 weeks
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg | Placebo
Number analyzed (Participants) | 67 | 66 | 67 | 71
Ratio
  Visit 2 (Day 8): number analyzed (Participants) | 66 | 61 | 62 | 70
  Visit 2 (Day 8) | -0.0003 (0.02279) | 0.0014 (0.01945) | -0.0016 (0.03487) | -0.0029 (0.02374)
  Visit 3 (Week 4): number analyzed (Participants) | 65 | 62 | 62 | 66
  Visit 3 (Week 4) | 0.0036 (0.01855) | 0.0024 (0.02095) | 0.0067 (0.02997) | -0.0024 (0.02539)
  Visit 4 (Week 8): number analyzed (Participants) | 61 | 61 | 58 | 65
  Visit 4 (Week 8) | 0.0151 (0.02153) | 0.0162 (0.02709) | 0.0258 (0.03233) | -0.0041 (0.02383)
  Visit 5 (Week 12): number analyzed (Participants) | 57 | 55 | 53 | 62
  Visit 5 (Week 12) | 0.0153 (0.02419) | 0.0175 (0.02270) | 0.0256 (0.02906) | -0.0082 (0.02882)
  Visit 6 (Week 16): number analyzed (Participants) | 54 | 50 | 52 | 56
  Visit 6 (Week 16) | 0.0142 (0.02195) | 0.0233 (0.02408) | 0.0229 (0.03260) | -0.0079 (0.02533)
  Visit 7 (Week 20): number analyzed (Participants) | 53 | 45 | 46 | 55
  Visit 7 (Week 20) | 0.0195 (0.02545) | 0.0192 (0.02672) | 0.0187 (0.03222) | -0.0063 (0.03037)
  Visit 8 (Week 24): number analyzed (Participants) | 50 | 41 | 41 | 54
  Visit 8 (Week 24) | 0.0171 (0.02612) | 0.0159 (0.02621) | 0.0216 (0.02587) | -0.0032 (0.02884)

11. Other Pre Specified Outcome: Mean (SD) Change From Baseline in Dual Energy X-ray Absorptiometry (DEXA) Scan T-score by Location at Week 24.
Description: Summary of DEXA Scan T-score at Visit 8 (Week 24) in the hip, femoral neck, and lumber spine. DEXA T-score was calculated based on actual measured bone density value and compared to a standard reference range for healthy young adult men.
  A bone density scan compares bone density with the bone density expected for a young healthy adult or a healthy adult of the same age, gender and ethnicity. The difference is calculated as a standard deviation (SD) score. The measures between the bone density and the expected value of a young healthy adult is known as the T score.
  The World Health Organization (WHO) classifies T scores as follows:
  * above -1 SD is normal
  * between -1 and -2.5 SD is defined as mildly reduced bone mineral density (BMD) compared with peak bone mass (PBM)
  * at or below -2.5 SD is defined as osteoporosis
Time Frame: Screening to Week 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg | Placebo
Number analyzed (Participants) | 67 | 66 | 67 | 71
T-score
  Hip: number analyzed (Participants) | 34 | 30 | 32 | 30
  Hip | 0.01 (0.382) | 0.05 (0.315) | -0.02 (0.323) | 0.01 (0.266)
  Femoral neck: number analyzed (Participants) | 34 | 30 | 32 | 31
  Femoral neck | -0.16 (0.337) | 0.02 (0.441) | -0.11 (0.392) | 0.03 (0.212)
  Lumber spine: number analyzed (Participants) | 34 | 28 | 31 | 30
  Lumber spine | -0.12 (0.279) | -0.08 (0.381) | -0.22 (0.351) | 0.07 (0.346)

12. Other Pre Specified Outcome: Mean (SD) Change From Baseline in DEXA Scan Density by Location at Week 24
Description: Summary of DEXA scan density at Visit 8 (Week 24) in the hip, femoral neck, and lumber spine. Bone density was evaluated with standard procedure for Hologic and General Electric Lunar scanners.
Time Frame: Screening to Week 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg | Placebo
Number analyzed (Participants) | 67 | 66 | 67 | 71
g/cm^2
  Hip: number analyzed (Participants) | 36 | 30 | 33 | 31
  Hip | -0.0026 (0.03990) | -0.0020 (0.03828) | -0.0072 (0.02724) | 0.0005 (0.03315)
  Femoral neck: number analyzed (Participants) | 35 | 30 | 33 | 31
  Femoral neck | -0.0248 (0.04583) | -0.0044 (0.06666) | -0.0116 (0.05139) | 0.0028 (0.02747)
  Lumber spine: number analyzed (Participants) | 36 | 29 | 32 | 31
  Lumber spine | -0.0167 (0.03174) | -0.0177 (0.05018) | -0.0255 (0.04044) | 0.0100 (0.04016)

13. Other Pre Specified Outcome: Mean (SD) Change From Baseline in Bone Turnover Markers by Parameter at Week 24.
Description: Descriptive statistics were presented for the following bone turnover marker parameters: type I collagen C-telopeptides, procollagen 1 N-terminal propeptide, osteocalcin, and bone specific alkaline phosphatase.
Time Frame: Screening to Week 24
Population: ITT Population. Discrepancies in numbers from the progress flow are due to missing samples either at baseline or wk 24/EOT.
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg | Placebo
Number analyzed (Participants) | 67 | 65 | 67 | 71
ug/L
  Type I Collagen C-Telopeptides: number analyzed (Participants) | 58 | 51 | 56 | 55
  Type I Collagen C-Telopeptides | 0.054 (0.1454) | 0.069 (0.1618) | 0.047 (0.1342) | 0.020 (0.2087)
  Procollagen 1 N-Terminal Propeptide: number analyzed (Participants) | 58 | 51 | 55 | 54
  Procollagen 1 N-Terminal Propeptide | 5.2 (8.31) | 5.0 (11.93) | 4.3 (11.68) | 1.8 (11.61)
  Osteocalcin: number analyzed (Participants) | 59 | 51 | 56 | 52
  Osteocalcin | 0.72 (2.891) | 0.35 (3.801) | 0.36 (3.604) | 0.30 (3.267)

14. Other Pre Specified Outcome: Change From Baseline in Bone Specific Alkaline Phosphatase at Week 24.
Description: Change from baseline in bone specific alkaline phosphatase at week 24 measured in U/L
Time Frame: 24 weeks
Population: ITT population on all available samples and including all wk 24 and end-of-treatment visit data.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg | Placebo
Number analyzed (Participants) | 58 | 51 | 56 | 55
U/L | 0.15 (3.187) | 0.69 (4.556) | 0.03 (3.629) | 0.29 (3.197)

ADVERSE EVENTS:
Time Frame: After randomisation and up to 90 days after the last administration of study drug.
Description: The following variables were recorded for each AE: verbatim/AE description and date for AE start and stop, severity, seriousness, causality rating, whether or not the AE caused the subject to discontinue, and the outcome. If the severity of the AE changed, a new AE had to be recorded. All ongoing AEs/SAEs were followed up until resolution or stabilisation or the last visit if in the Investigator's opinion, the AE was unlikely to resolve due to the subject's underlying disease.
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/66 | 0/67 | 0/71
Serious Adverse Events (participants affected / at risk) | 2/67 | 2/66 | 5/67 | 5/71
Other Adverse Events (participants affected / at risk) | 37/67 | 39/66 | 47/67 | 41/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BGS649 0.1 mg (N=67) | BGS649 0.3 mg (N=66) | BGS649 1.0 mg (N=67) | Placebo (N=71)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthritis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BGS649 0.1 mg (N=67) | BGS649 0.3 mg (N=66) | BGS649 1.0 mg (N=67) | Placebo (N=71)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 3 (4) | 2 (2) | 5 (5)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bacterial prostatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematocrit increased (Investigations) | 1 (2) | 4 (5) | 5 (6) | 0 (0)
Prostatic specific antigen increased (Investigations) | 2 (2) | 1 (1) | 4 (4) | 2 (2)
Blood triglycerides increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Weight increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood insulin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood prolactin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heart rate irregular (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Low density lipoprotein increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 7 (8) | 3 (4) | 4 (4) | 2 (3)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Central nervous system lesion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Complex regional pain syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Primary headache associated with sexual activity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sensory loss (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 4 (4) | 1 (1) | 2 (2)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cyst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Energy increased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Libido decreased (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Apathy (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Euphoric mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Loss of libido (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypochloraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Androgenetic alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Penile ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bladder outlet obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glycosuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erection increased (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatic mass (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spontaneous penile erection (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Testicular hypertrophy (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 2 (2) | 5 (5) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polycythaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cyanosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/69/NCT02730169/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-07): https://cdn.clinicaltrials.gov/large-docs/69/NCT02730169/SAP_001.pdf